CLINICAL TRIAL: NCT05634174
Title: Identifying Responsible Signaling Pathway for Adrenergic Beta-3 Receptor Regulation in Human Subcutaneous White Adipose Tissue
Brief Title: ADRB3 Signaling Pathway in Human Adipose Tissue
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Vala Hamidi, Assistant Clinical Professor, University of California, San Diego, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UC-MEDVH-01
Record Dates: First submitted 2022-11-21; First posted 2022-12-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Prediabetes
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Obese Group (Experimental): Single dose, 100mg oral mirabegron in Obese Insulin Resistant adults
  Interventions: Drug: Mirabegron
- Non-Obese Group (Experimental): Single dose, 100mg oral mirabegron in Non-Obese adults
  Interventions: Drug: Mirabegron

INTERVENTIONS:
Drug: Mirabegron — Single dose, 100mg oral mirabegron
  Other Names: Myrbetriq

SUMMARY:
This study will examine the gene expression of the adrenergic Beta-3 receptor (ADRB3) regulation in human subcutaneous adipose tissue before and after treatment with mirabegron, an ADRB3 agonist. Gene expression will be compared across two groups, lean and obese participants. There will be a total of three study visits: Screening/Eligibility, Pre-Dose Adipose Tissue Biopsy and Post-Dose Adipose Tissue Biopsy. Participants will be given a single dose of 100mg oral mirabegron on the day of the Post-Dose Adipose Tissue Biopsy.The trial design is a single-center, phase 1, open-label, exploratory study to examine the adipocyte gene expression in adults treated with 1 dose of 100mg oral mirabegron.

DETAILED DESCRIPTION:
The trial design is a single-center, phase 1, open-label, exploratory study to examine the adipocyte gene expression in adults treated with 1 dose of 100mg oral mirabegron.

This is an exploratory study to examine the effects of a single dose of mirabegron on adipocytes in insulin resistant obese individuals and lean controls. Approximately 40 patients over the age of 18 will be recruited for the study (20 obese individuals with insulin resistance and 20 lean controls).

There will be a total of three study visits: Screening/Eligibility, Pre-Dose Adipose Tissue Biopsy and Post-Dose Adipose Tissue Biopsy. All visits will take place at the ACTRI research clinic at UC San Diego. The Screening/Eligibility visit will involve collection of safety data and eligibility criteria, medical/medication history, physical exam, vitals, ECG and collection of urine and blood for safety laboratory analysis. The procedures completed at the Pre-Dose visit will be, vitals, re-review of medical history and changes since last visit, indirect calorimetry, an oral glucose tolerance test (OGTT), an adipose tissue biopsy, blood sample collection and study drug dispensing (one dose to be taken the morning of the following visit). The procedures completed at the Post-Dosing visit will be identical to those completed at the Baseline visit, except there will not be an OGTT at the Post-Dosing Visit.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provision of signed and dated informed consent form 2. Stated willingness to comply with all study procedures and availability for the duration of the study 3. Males and females 18-70 years old 4. Lean participants, defined as:

  * BMI <27 kg/m2
  * Normal glucose tolerance defined as fasting glucose less than 100 mg/dL or HbA1c of less than 5.7% at the time of the screening visit 5. Obese Insulin resistant participants, defined as:
  * BMI 30-40 kg/m2
  * Prediabetes defined as fasting glucose levels of 100 to 125 mg/dL or HbA1c of 5.7% to 6.4%
  * Agreement to adhere to Lifestyle Considerations (see section 5.3) throughout study duration

Exclusion Criteria:

* 1. Diabetes, defined as fasting glucose ≥ 126 mg/dL, HbA1c ≥ 6.5%, or diagnosis of diabetes 2. Pregnancy or lactation 3. Currently taking therapeutic anticoagulation which might increase risk of bleeding from fat biopsy (e.g., warfarin, direct oral anticoagulants) 4. History of eating disorder 5. Currently enrolled in a weight-loss or weight-management program 6. On a special or prescribed diet for other reasons (e.g., Celiac disease) 7. Currently taking any medication that is meant for, or has known effect on, appetite 8. Any history of surgical intervention for weight management 9. Abnormal screening labs (renal dysfunction (eGFR < 30 ml/min/1.73 m2), anemia, hypo- or hyperthyroidism, coagulopathy, abnormal liver function (AST, ALT > 3x upper limit of normal) 10. Local or systemic infectious disease with fever or requiring antibiotic within four weeks of screening visit 11. QTc interval above normal or the current use of any concomitant QT-prolonging drug 12. A clinically significant abnormal ECG 13. Current addiction to alcohol or substances of abuse 14. Unwillingness or language barriers precluding adequate understanding or cooperation 15. Use of systemic corticosteroids or other medication known to cause insulin resistance in previous six weeks prior to the screening visit and throughout the study 16. Diagnosis of bladder outlet obstruction or use of antimuscarinic medications for treatment of overactive bladder 17. Use of β-adrenergic receptor blockers or calcium channel blockers 18. Heart disease including Coronary Artery Disease (CAD), Congestive Heart Failure (CHF), or cardiac arrhythmias 19. Uncontrolled sever hypertension (Defined as systolic blood pressure ≥ 180 mm Hg and/or diastolic blood pressure ≥110 mm Hg) 20. Any other condition(s) that might reduce the chance of obtaining study data, or that might cause safety concerns, or that might compromise the ability to give truly informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
ADRB3 gene expression | 28 days (± 14 days)
  The change from baseline in ADRB3 gene expression as measured by qPCR
ADRB3 protein levels | 28 days (± 14 days)
  The change from baseline in ADRB3 protein levels as measured by Western Blot
Glycerol Measured Catecholamine Sensitivity | 28 days (± 14 days)
  The change from baseline in catecholamine sensitivity as measured by glycerol from adipose tissue lipolysis
Free Fatty Acid measured Catecholamine Sensitivity | 28 days (± 14 days)
  The change from baseline in catecholamine sensitivity as measured by Free Fatty Acid from adipose tissue lipolysis

SECONDARY OUTCOMES:
FGF-21 Adipokine Gene Expression | 28 days (± 14 days)
  The change from baseline in FGF-21 gene expression as measured by qPCR
IL-6 Adipokine Gene Expression | 28 days (± 14 days)
  The change from baseline in IL-6 gene expression as measured by qPCR

OTHER OUTCOMES:
ADRB3 Signaling Pathway | 28 days (± 14 days)
  Identification of ADRB3 signaling pathway as measured by RNA sequencing of adipocytes

CONTACTS AND LOCATIONS:
Locations (1):
- UC San Diego Altman Clinical & Translational Research Institute, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No